CLINICAL TRIAL: NCT00694265
Title: Sonographic Follow-up of Patients With Carpal Tunnel Syndrome Undergoing Surgical or Conservative Treatment: Prospective Cohort Study.
Brief Title: Sonographic Follow-up of Patients With Carpal Tunnel Syndrome Undergoing Surgical or Conservative Treatment
Acronym: CTS
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Peter Jüni, MD, Institute of Social and Preventive Medicine, University of Bern, Switzerland
Other Study IDs: CTU_CTS; UBern_CTS
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Median Nerve; Ultrasonography; Prospective cohort study
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Decompression; Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Surgical treatment
  Interventions: Procedure: Decompression
- 2: Conservative treatment
  Interventions: Procedure: Conservative treatment

INTERVENTIONS:
Procedure: Decompression — Surgical decompression of the median nerve
  Groups: 1
Procedure: Conservative treatment — Conservative treatment typically consisted of splinting and corticosteroid injections
  Groups: 2

SUMMARY:
In wrists with carpal tunnel syndrome (CTS) the sonographically measured largest cross-sectional area (CSA) of the median nerve is increased. We compared the changes in largest CSA in wrists undergoing surgical decompression and wrists undergoing conservative treatment of CTS.

DETAILED DESCRIPTION:
Objective:

In wrists with carpal tunnel syndrome (CTS) the sonographically measured largest cross-sectional area (CSA) of the median nerve is increased. We compared the changes in largest CSA in wrists undergoing surgical decompression and wrists undergoing conservative treatment of CTS.

Methods:

Prospective cohort study in 55 consecutive patients with 78 wrists with established CTS, including 60 wrists with surgical decompression and 18 wrists with conservative treatment. A sonographic examination was scheduled before and at 4 months after initiation of treatment. Changes in CSA between wrists with surgical and wrists with conservative treatment were compared using linear regression models.

ELIGIBILITY:
Inclusion Criteria:

* wrists with established CTS

Exclusion Criteria:

* prior surgery for CTS
* traumatic lesions
* coexistent neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected CTS
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2002-01; Primary Completion 2003-06 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Measure of the largest cross-sectional area (CSA) of the median nerve | Before and 4 months after initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jüni, MD, Study Director — Institute of Social and Preventive Medicine, University of Bern, Switzerland; Hans-Rudolf Ziswiler, MD, Principal Investigator — Dep. of Rheumatology, Immunology and Allergology, Bern University Hospital, Switzerland
Locations (1):
- Dep. of Plastic and Hand Surgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Ziswiler HR, Reichenbach S, Vogelin E, Bachmann LM, Villiger PM, Juni P. Diagnostic value of sonography in patients with suspected carpal tunnel syndrome: a prospective study. Arthritis Rheum. 2005 Jan;52(1):304-11. doi: 10.1002/art.20723. PMID 15641050
- [Background] Bachmann LM, Juni P, Reichenbach S, Ziswiler HR, Kessels AG, Vogelin E. Consequences of different diagnostic "gold standards" in test accuracy research: Carpal Tunnel Syndrome as an example. Int J Epidemiol. 2005 Aug;34(4):953-5. doi: 10.1093/ije/dyi105. Epub 2005 May 23. PMID 15911545